CLINICAL TRIAL: NCT03476278
Title: Evaluation of Factors Associated With Patient Satisfaction and Mood-State in Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hande G. Aytuluk, Principal Investigator, Derince Training and Research Hospital
Other Study IDs: U1111-1211-0907
Record Dates: First submitted 2018-03-17; First posted 2018-03-26 (Actual); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Outcome Assessment; Patient Satisfaction
Keywords: Outcome Assessment (Health Care); Patient Satisfaction; Perioperative Period; Regional Anesthesia; Surveys and Questionnaires
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- regional, questionnaire: patients who underwent surgery under regional anesthesia.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Postoperative questionnaire, and records of complications in the peri-operative period

SUMMARY:
Patient satisfaction is an important subjective measure of healthcare quality which contributes to evaluation of the structure, process and outcome of services. The key factor in patient satisfaction is adequate perioperative information of the patient and communication between healthcare providers and patient or patient's kin.

There are few studies in anesthesia that have assessed patient satisfaction and mood-state during regional anesthesia.

The investigators aimed to evaluate factors associated with patient satisfaction from regional anesthesia procedure and mood-state of patients who underwent surgery under regional anesthesia.

DETAILED DESCRIPTION:
Patient satisfaction is an important subjective measure of healthcare quality which contributes to evaluation of the structure, process and outcome of services. Many factors contribute to patient satisfaction, including institutional structure, interpersonal relationships, and a patient' expectations. Age, gender, social insurance, educational and social statue also play role in patient satisfaction. The key factor in patient satisfaction is adequate perioperative information of the patient and communication between healthcare providers and patient or patient's kin.

The success of regional anesthesia is influenced by several factors. Most patients expect uneventful perioperative process. Nevertheless, recovery from surgery and anesthesia is sometimes complicated by major and minor complaints including pain, nausea, vomiting and other. Although there is no scientific or clinical evidence that regional anesthesia is superior to general anesthesia, regional anesthesia has some advantages like keeping consciousness of the patient during surgery, continuation of spontaneous breathing, avoiding the loss of protective reflexes, allowing early mobilization in the postoperative period and shortening the length of hospital stay. However, the major contraindication for regional anesthesia is the patient's unwillingness.

There are few studies in anesthesia that have assessed patient satisfaction and mood-state during regional anesthesia.

The investigators aimed to evaluate factors associated with patient satisfaction from regional anesthesia procedure and mood-state of patients who underwent surgery under regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

- patients who underwent gynecological and obstetrical, urological, orthopedic and general surgical procedures under general anesthesia

Exclusion Criteria:

- clinically significant psychiatrically ill illiterate patients who received general anesthesia patients that have speech, hearing, or understanding problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent gynecological and obstetrical, urological, orthopedic and general surgical procedures under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2011-01-01 (Actual); Study Completion 2011-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vildan Akpinar, MD, Study Director — Izmir Bozyaka Training and Research Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The investigators do not prefer to share the study plan and records.

REFERENCES:
- [Result] De Andres J, Valia JC, Gil A, Bolinches R. Predictors of patient satisfaction with regional anesthesia. Reg Anesth. 1995 Nov-Dec;20(6):498-505. PMID 8608068
- [Result] Donabedian A. Evaluating the quality of medical care. 1966. Milbank Q. 2005;83(4):691-729. doi: 10.1111/j.1468-0009.2005.00397.x. No abstract available. PMID 16279964
- [Result] Lohr KN, Donaldson MS, Harris-Wehling J. Medicare: a strategy for quality assurance, V: Quality of care in a changing health care environment. QRB Qual Rev Bull. 1992 Apr;18(4):120-6. doi: 10.1016/s0097-5990(16)30518-8. PMID 1630793
- [Result] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Result] Hall JA, Dornan MC. Patient sociodemographic characteristics as predictors of satisfaction with medical care: a meta-analysis. Soc Sci Med. 1990;30(7):811-8. doi: 10.1016/0277-9536(90)90205-7. PMID 2138357
- [Derived] Tosuner Akpinar V, Koroglu L, Gurbuz Aytuluk H. Evaluation of factors associated with patient satisfaction and mood-state in regional anesthesia. Agri. 2019 Apr;31(2):57-62. doi: 10.5505/agri.2018.71363. PMID 30995331

RESULTS

PARTICIPANT FLOW:
Groups:
- Regional: patients who underwent surgery under regional anesthesia.
  Questionnaire: Postoperative questionnaire, and records of complications in the peri-operative period
Period: Overall Study
Arm/Group | Regional
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regional
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 274
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 192
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Patient Satisfaction
Description: satisfaction of patients during regional anesthesia (patients will be handed a questionnaire about their satisfaction in recovery room or in ward. They will be able to mark only one option: satisfaction, dissatisfaction)
Time Frame: 1 day (peri-operative)
Measure: Count of Participants; unit: Participants
Groups:
- Satisfaction: satisfied patients who underwent surgery under regional anesthesia.
  Questionnaire: Postoperative questionnaire, and records of complications in the peri-operative period
- Dissatisfaction: dissatisfied patients who underwent surgery under regional anesthesia.
  Questionnaire: Postoperative questionnaire, and records of complications in the peri-operative period
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 300 | 300
Participants | 247 | 53

2. Primary Outcome: Overall Mood-state
Description: mood-state of patients during regional anesthesia (patients will be handed a questionnaire about their mood-state in recovery room or in ward. They will be able to mark more than one option about their mood-state: safe, unsafe, comfortable, exited, anxious)
Time Frame: 1 day
Population: Patients were able to mark more than one option in the part of the questionnaire about mood-state: safe, unsafe, comfortable, exited, anxious. If patient was heavily sedated and too confused to participate, the questionnaire was handed at the ward after recovery.
Measure: Count of Participants; unit: Participants
Groups:
- Safe: Patients who feel safe under regional anesthesia
- Unsafe: Patients who feel unsafe under regional anesthesia
- Comfortable: Patients who feel comfortable under regional anesthesia
- Excited: Patients who feel excited under regional anesthesia
- Anxious: Patients who feel anxious under regional anesthesia
Arm/Group | Safe | Unsafe | Comfortable | Excited | Anxious
Number analyzed (Participants) | 300 | 300 | 300 | 300 | 300
Participants | 137 | 20 | 109 | 115 | 67

3. Secondary Outcome: Patient Satisfaction According to Age
Description: patient satisfaction according to age under regional anesthesia
Time Frame: 1 day (postoperative)
Measure: Count of Participants; unit: Participants
Groups:
- Satisfaction; Dissatisfaction: patients who underwent surgery under regional anesthesia.
  Questionnaire: Postoperative questionnaire, and records of complications in the peri-operative period
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Participants
  18-25 | 23 | 1
  26-35 | 30 | 16
  36-45 | 77 | 12
  46-55 | 54 | 10
  56-65 | 41 | 10
  66-75 | 22 | 4

4. Secondary Outcome: Patient Satisfaction According to Gender
Description: patient satisfaction according to gender under regional anesthesia
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Satisfaction: satisfied patients who underwent surgery under regional anesthesia.
  Patients were only able to mark one option: satisfied or dissatisfied.
- Dissatisfaction: dissatisfied patients who underwent surgery under regional anesthesia.
  Patients were only able to mark one option: satisfied or dissatisfied.
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Participants
  Female | 83 | 25
  Male | 164 | 28

5. Secondary Outcome: Patient Satisfaction According to Education
Description: patient satisfaction from regional anesthesia according to their highest level of education received.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Participants
  Primary school | 112 | 24
  Junior high school | 32 | 8
  High school | 59 | 15
  University | 44 | 6

6. Secondary Outcome: Patient Satisfaction According to the Type of Surgery
Description: patient satisfaction according to the type of surgery under regional anesthesia
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Participants
  General | 56 | 16
  Orthopedic | 51 | 9
  Gynecology & obstetric | 38 | 16
  Urology | 102 | 12

7. Secondary Outcome: Patient Satisfaction According to Past Regional Anesthesia Experience
Description: patient satisfaction according to past regional anesthesia experience under regional anesthesia
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Participants
  yes | 115 | 15
  no | 132 | 38

8. Secondary Outcome: Patient Satisfaction According to Preoperative Information
Description: Patients who were given additional preoperative information about regional anesthesia and the things they would encounter during regional anesthesia (ie: they will feel the touches but pain is not expected to be felt, they can feel nausea because of the side-effect of the regional block, what will be done if the regional blocks are unsuccessful and they feel pain,..etc.)
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Participants
  yes | 241 | 44
  no | 6 | 9

9. Secondary Outcome: Patient Satisfaction According to Intra-operative Adverse Events
Description: patient satisfaction according to intra-operative adverse events under regional anesthesia
Time Frame: 1 day
Measure: Number; unit: number of experienced adverse events
Units Other Than Participants: adverse events
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Number analyzed (adverse events) | 123 | 37
number of experienced adverse events
  Hypotension | 61 | 11
  Bradycardia | 22 | 5
  Nausea-vomiting | 36 | 12
  Pain | 4 | 9

10. Secondary Outcome: Patient Satisfaction According to Recovery Room Adverse Events
Description: patient satisfaction according to recovery room adverse events following surgery under regional anesthesia
Time Frame: 1 day
Measure: Count of Units; unit: adverse events
Units Other Than Participants: adverse events
Arm/Group | Satisfaction | Dissatisfaction
Number analyzed (Participants) | 247 | 53
Number analyzed (adverse events) | 98 | 19
adverse events
  Hypotension | 26 | 4
  Bradycardia | 30 | 6
  Nausea-vomiting | 14 | 5
  Pain | 28 | 4

11. Secondary Outcome: Mood State According to Age
Description: Patients' mood state according to age
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Safe | Unsafe | Comfortable | Excited | Anxious
Number analyzed (Participants) | 137 | 20 | 109 | 115 | 67
Participants
  18-25 | 6 | 0 | 8 | 12 | 5
  26-35 | 16 | 5 | 11 | 26 | 16
  36-45 | 42 | 5 | 32 | 34 | 22
  46-55 | 36 | 5 | 24 | 19 | 10
  56-65 | 24 | 3 | 24 | 17 | 10
  66-75 | 13 | 2 | 10 | 7 | 4

12. Secondary Outcome: Mood State According to Gender
Description: Patients' mood state according to gender
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Safe | Unsafe | Comfortable | Excited | Anxious
Number analyzed (Participants) | 137 | 20 | 109 | 115 | 67
Participants
  Female | 45 | 8 | 33 | 48 | 28
  Male | 92 | 12 | 76 | 67 | 39

13. Secondary Outcome: Mood State According to Education
Description: Patients' mood state according to their highest degree of education received
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Safe | Unsafe | Comfortable | Excited | Anxious
Number analyzed (Participants) | 137 | 20 | 109 | 115 | 67
Participants
  Primary school | 64 | 10 | 57 | 47 | 32
  Junior high school | 16 | 1 | 15 | 15 | 11
  High school | 31 | 7 | 21 | 37 | 14
  University | 26 | 2 | 16 | 16 | 10

14. Secondary Outcome: Mood State According to Preoperative Information
Description: as for outcome 8
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Safe | Unsafe | Comfortable | Excited | Anxious
Number analyzed (Participants) | 137 | 20 | 109 | 115 | 67
Participants
  yes | 134 | 17 | 106 | 110 | 60
  no | 3 | 3 | 3 | 5 | 7

ADVERSE EVENTS:
Time Frame: 1 day
Description: adverse events (ie: bradycardia, hypotension, nausea-vomiting, pain) due to regional anesthesia were collected. However these events were not related to the participant's participation in the research (this research is a questionnaire).
Arm/Group | Regional, Questionnaire
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 85/300
Other Adverse Events (participants affected / at risk) | 0/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regional, Questionnaire (N=300)
Bradycardia (Cardiac disorders) | 32 (32)
hypotension (Cardiac disorders) | 83 (83)
nausea-vomitting (Gastrointestinal disorders) | 24 (24)
pain (Surgical and medical procedures) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT03476278/Prot_SAP_000.pdf